CLINICAL TRIAL: NCT01328483
Title: Role of Intrapartum Oropharyngeal (IP-OP) Suction in Neonates Born Through Meconium Stained Amniotic Fluid on Meconium Aspiration Syndrome
Brief Title: Effect Of Intrapartum Oropharyngeal (IP-OP) Suction on Meconium Aspiration Syndrome
Acronym: MSAF-OPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Professor, Department of Neonatology, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LHMC/21/2008/MSAF-OPS
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Meconium Aspiration Syndrome
Keywords: Neonates; Intrapartum Oropharyngeal Suctioning; Meconium Aspiration Syndrome
MeSH Terms: conditions — Meconium Aspiration Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Intrapartum Oropharyngeal (IP-OP) Suction (No Intervention): Neonates randomized to No IP-OP group received supportive treatment as per standard unit protocols. They were also assessed as vigorous or non-vigorous and received care according to NRP 2005.
- Intrapartum Oropharyngeal (IP-OP) suction (Experimental): The neonates randomized to IP-OP group were provided oropharyngeal suctioning at the delivery of head before the delivery of shoulder, using suction machine at a negative pressure of 100mm of Hg or Dee Lee's suction trap in the event of electricity failure or non availability of suction machine.Subsequently, all the neonates born through MSAF were assessed by pediatrician as vigorous or non vigorous and provided care as per NRP guidelines 2005.
  Interventions: Procedure: Intrapartum Oropharyngeal Suctioning

INTERVENTIONS:
Procedure: Intrapartum Oropharyngeal Suctioning — After delivery of the head, the infant's mouth and nose were suctioned. Nose was suctioned after the mouth and throat. Oropharyngeal suctioning was performed using a 10 french suction catheter with suction pressure of 100mm Hg or De Lee's suction trap in event of electricity failure or non availability of suction machine
  Arms: Intrapartum Oropharyngeal (IP-OP) suction

SUMMARY:
The purpose of the study is to evaluate the role of routine suctioning of the oropharynx before the delivery of shoulders in preventing breathing difficulty and subsequent lung disease in babies born through meconium stained amniotic fluid. Normally babies do not pass meconium while in utero. In response to hypoxic stress babies may pass meconium before birth and are likely to be candidates for problems related to meconium passage and its inhalation leading to meconium aspiration syndrome(MAS). It is believed that clearing the airways of meconium at the time of birth can decrease the risk of MAS. It had been a routine practice to suction the mouth, pharynx and nose of the baby as soon as the head of the infant is delivered prior to delivery of the shoulders followed by tracheal intubation and suction in babies with poor breathing efforts to clear the airways of the meconium. however recent studies have shown the futility of this procedure in preventing MAS along with an increased risk of complications to baby due to suctioning. In view of the uncertainty regarding the effectiveness of this procedure in a resource poor country, the investigators decided to evaluate the effect of intrapartum-oropharyngeal suction in preventing or decreasing the incidence of MAS in such babies.

DETAILED DESCRIPTION:
Meconium passage in newborn infants is a developmentally programmed event normally occurring within first 24-48 hours of birth. Intra uterine meconium passage in near term or term fetuses has been associated with feto-maternal stress factors and/or infections, whereas meconium passage in post term pregnancies has been attributed to gastro-intestinal maturity. Meconium staining of amniotic fluid occurs in 12% of all live births per annuum. Aspiration of meconium that occurs during intra uterine life or after delivery with the first few breaths may result in or contribute to respiratory pathology known as meconium aspiration syndrome (MAS) which represents a leading cause of perinatal morbidity, occurring in 5-20% of all babies born through MSAF.

Several studies have shown that by clearing the airways of meconium at the time of birth, meconium aspiration pneumonia can be virtually eliminated. Based on these results, the American Heart Association and American Academy of Pediatrics had recommended a combined obstetric and pediatric approach to the infant with MSAF in the year 2000. As per this approach infants mouth, pharynx and nose were to be suctioned as soon as the head of the infant is delivered prior to delivery of the shoulders using a 10 french catheter followed by tracheal intubation and suction in non-vigorous infants to clear the airways of the meconium.

Accumulating evidence in the form of a large RCT from developed world has shown the futility of intrapartum-oropharyngeal suction leading to, omission of this procedure from resuscitation guidelines published in the year 2005.

Even though International Liaison Committee on Resuscitation recommends no need for IP- OP suction based on a single RCT conducted in a developed world with universal institutional deliveries and strict fetal surveillance, the same may not be true in set ups with unbooked and late second stage arrivals of the mother with prolonged fetal distress and virtually no perinatal surveillance.

Hence the purpose of this randomized controlled trial is to evaluate the effectiveness of intrapartum-oropharyngeal suction in preventing or decreasing the incidence of MAS in term neonates born through MSAF in resource poor setting in a developing country.

ELIGIBILITY:
Inclusion Criteria:

* Gestation >/= 37 weeks
* Meconium staining of amniotic fluid
* Cephalic presentation
* Singleton pregnancy

Exclusion Criteria:

* Babies with major congenital malformations (if known antenatally)
* Hydrops fetalis
* Refusal of consent
* Chromosomal anomalies

Max Age: 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 540 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Meconium Aspiration Syndrome | First 72 hours of life or till discharge
  Occurrence of Meconium aspiration syndrome as assessed by (all of these)
  * Birth through Meconium Stained Amniotic Fluid,
  * Presence of respiratory distress (as defined as RR>60/min, Subcostal retractions or Intercostal Retractions or Grunt)
  * Need for supplemental oxygen to maintain oxygen saturation > 92%
  * Need for supplemental oxygen by two hours of life and continued beyond 12 hours of life
  * Presence of radiological features of MAS on X-ray chest

SECONDARY OUTCOMES:
Mortality | First 72 hours of life or till discharge
Severity of MAS | First 72 hours of life or till discharge
  Severity of MAS was defined as:
  1. Mild MAS: oxygen requirement <40% and for <48 Hours
  2. Moderate MAS: Oxygen requirement of >40% for any duration or oxygen requirement of <40% for>48 hours or need for CPAP
  3. Severe MAS: need for mechanical ventilation
Duration of hospital stay | First 72 hours of life or till discharge
Respiratory Support | First 72 hours of life or till discharge
  1. Requirement of respiratory support
  2. The mode of respiratory support viz. Supplemental Oxygen therapy, CPAP, Mechanical ventilation, High Frequency ventilation
  3. Duration of each kind of respiratory support required
Incidence of air leaks | First 72 hours of life or till discharge
  Pneumothorax as seen by transillumination and confirmed by Chest Xray

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MBBS, MD, DM, Principal Investigator — Lady Hardinge Medical College, New Delhi, India
Locations (1):
- Kalawati Saran children's Hospital, Lady Hardinge Medical College, New Delhi, New delhi, India

REFERENCES:
- [Derived] Nangia S, Pal MM, Saili A, Gupta U. Effect of intrapartum oropharyngeal (IP-OP) suction on meconium aspiration syndrome (MAS) in developing country: A RCT. Resuscitation. 2015 Dec;97:83-7. doi: 10.1016/j.resuscitation.2015.09.394. Epub 2015 Oct 11. PMID 26449871